CLINICAL TRIAL: NCT06248398
Title: Impact of Robotic Cochlear Implantation on Hearing Performance in Noise
Acronym: ROBOT-IC-BRUIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: APHP211330; 2023-A00837-38 (Other: N°IDRCB)
Record Dates: First submitted 2023-12-08; First posted 2024-02-08 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Severe to Profound Hearing Loss
Keywords: Cochlear implant; Manual insertion; Robotic assistance insertion; Hearing understanding in noise; Quality of life
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Patient having cochlear implantation surgery with RobOtol®.
  Interventions: Procedure: Surgery with RobOtol®
- Control arm (Other): Patient having conventional manual cochlear implantation surgery.
  Interventions: Procedure: Conventional manual surgery

INTERVENTIONS:
Procedure: Surgery with RobOtol® — Patient having cochlear implantation surgery with RobOtol®.
  Arms: Experimental arm
Procedure: Conventional manual surgery — Patient having conventional manual cochlear implantation surgery
  Arms: Control arm

SUMMARY:
The purpose of this study is to compare two methods of cochlear implantation : conventional manual insertion versus robot-assisted in order to verify whether robotic insertion provides better performance in the noisy environment.

To do this, we will compare the two methods of insertion of the electrode holder, on 140 patients candidates for cochlear implantation randomized in two groups (70 conventional surgery versus 70 robot-assisted surgery). All patients will be recruited during 17 months, in our Ear, nose and throat (ENT) Department of the Pitié-Salpêtrière hospital group, the first center for adult patients established in France (on average 180 patients/year).

Patient will be followed for 9 months with clinical evaluation, imaging, audiometric, listening effort and quality of life assessments. These evaluations will be carried out preoperatively and postoperatively at 3 months and 6 months post-activation of the cochlear implant.

DETAILED DESCRIPTION:
In the case of severe (70 to 90dB loss) and profound (>90dB loss) hearing loss, when conventional hearing aids no longer provide sufficient benefit, cochlear implantation remains the only possible solution for hearing rehabilitation. In implanted patients, a clear improvement in communication in silence is observed, but almost all patients have difficulty understanding speech in noisy environments. Cochlear implantation involves inserting an electrode holder into the cochlea during a surgical procedure under general anesthesia. The insertion of the electrode holder must be as minimally traumatic as possible in order to preserve the cochlear structures and avoid post-operative fibrosis that could impact the auditory outcomes.

The conventional method of this surgery is the manual insertion of the electrode holder. In recent years, robotic assistance, the RobOtol®, has been developed with the aim of avoiding the jerks of the surgeon's hand and improving the precision of the insertion. RobOtol® has had its CE marking since 2016 and is used in several hospitals in France and abroad.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years old
* Patients with an indication for uni or bilateral, simultaneous or sequential cochlear implantation: severe to profound bilateral deafness with intelligibility ≤70% for Fournier dissyllabic words, in free field, at 60dB with adapted hearing aids.
* Patient able to understand the information note and give written consent
* Affiliation to a French social security system

Exclusion Criteria:

* Patient who does not speak French
* Etiologies of deafness known to be of bad prognosis (auditory neuropathy, congenital profound deafness, immediate post-meningitis profound deafness, vestibular schwannoma on the side of the ear to be implanted)
* Impossibility of testing the effect of the cochlear implant alone on hearing results (cochlear implantation in the context of unilateral deafness or fluctuating deafness)
* Cochlear implantation requiring the use of a perimodiolar electrode holder.
* Pregnant and breastfeeding women
* Patients wearing electronic devices, in direct connection with the brain or nervous system
* Patient included in another interventional study (Jardé 1)
* Patient under legal protection (guardianship or curatorship) or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Auditory performance in noise with the cochlear implant | At 6 months post-implantation
  Evolution of the intelligibility score (Variation of the percentage of words understood) for monosyllabic Lafon words presented at 60 dB SPL with a signal-to-noise ratio of 10 dB (SNR10) between the preoperative score and the score at 6 months post-implantation

SECONDARY OUTCOMES:
Hearing performance in noise after robotic cochlear implantation compared to conventional manual cochlear implantation for phonemes | At 3 and 6 months post-implantation
  Evolution of the intelligibility score (Variation of the percentage of words and phonemes understood) for monosyllabic Lafon words presented at 60 dB SPL with a signal-to-noise ratio of 10 dB (SNR10) between the preoperative score and the score at 3 months and at 6 months post-implantation.
Hearing performance in noise under ecological conditions after robotic cochlear implantation compared to conventional manual cochlear implantation | At 3 and 6 months post-implantation
  Evolution of the intelligibility score (Variation of the percentage of words understood) for Fr-Bio words presented at 60 dB SPL with a signal-to-noise ratio of 10 dB (SNR10) between the preoperative score and the score at 3 months and at 6 months post-implantation. The noise will be an ecological noise (restaurant or street noise) using the Immersion® system.
Hearing performance in silence after robotic cochlear implantation compared to conventional manual cochlear implantation for words | At 3 and 6 months post-implantation
  Evolution of the intelligibility score (Variation of the percentage of words understood) for monosyllabic Lafon words presented at 60 dB SPL in quiet between the preoperative score and the score at 3 months and at 6 months post-implantation.
Hearing performance in silence after robotic cochlear implantation compared to conventional manual cochlear implantation for phonemes | At 3 and 6 months post-implantation
  Evolution of the intelligibility score (Variation of the percentage of phonemes understood) for monosyllabic Lafon words presented at 60 dB SPL in quiet between the preoperative score and the score at 3 months and at 6 months post-implantation.
The subjective benefit on tinnitus after robotic cochlear implantation compared to conventional manual cochlear implantation | At 3 and 6 months post-implantation
  Evolution of the Patient's Related Outcomes Measures using questionnaire concerning the tinnitus with the Tinnitus Handicap Inventory (THI)
The subjective benefit on quality of life after robotic cochlear implantation compared to conventional manual cochlear implantation | At 3 and 6 months post-implantation
  Evolution of the Patient's Related Outcomes Measures using the questionnaire concerning the quality of life with the Cochlear Implant Quality of Life (CIQOL)
The position of the electrode array in the cochlea during manual and robotic insertions | At day one post -implantation
  the position of each electrode will be analyzed blindly on the post-operative CT-scan.
The impact of a translocation on auditory performance in silence and in noise | At 3 and 6 months post-implantation
  Auditory scores measured at 3 and 6 months after implantation will be correlated to the presence of a translocation of the electrode array assessed on the post-operative CT scan.
The effort of listening in silence and in noise after manual and robotic insertions assessed with the Speech, Spatial and Qualities of Hearing Scale (SSQ) | At 3 and 6 months post-implantation
  The effort of listening will be analyzed with SSQ scale
The effort of listening in silence and in noise after manual and robotic insertions assessed with a visual analog scale | At 3 and 6 months post-implantation
  The effort of listening will be analyzed after each audiologic test with a visual analog scale, using which the patient will rate from 0 to 10 the effort made to understand the words presented (Bräcker et al., 2019)
The preservation of residual hearing after cochlear implantation in cases with residual hearing before surgery | At 30 days, 3 months and 6 months post-implantation
  Evolution of auditory thresholds measured with tonal audiometry between preoperative and postoperative measurements on the operated ear.
The presence of postoperative vertigo in case of robotic cochlear implantation compared to manual implantation | At 7 days, 3 months and 6 months post-implantation
  Evaluation of vertigo with the Dizziness Handicap Inventory (DHI) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ghizlene LAHLOU, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.